CLINICAL TRIAL: NCT01348594
Title: The Impact of Vitamin D on Implantation and Clinical Pregnancy Rates Following in Vitro Fertilization
Brief Title: The Impact of Vitamin D Status on in Vitro Fertilization (IVF) Outcomes
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Kimberly Liu, Reproductive Endocrinology and Infertility Specialist, University of Toronto
Other Study IDs: 10-0288-E
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Vitamin D Status
Keywords: Vitamin D; In vitro Fertilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitamin D deficient
- Vitamin D sufficient

SUMMARY:
Infertility is a common and psychologically devastating problem for 20% of Canadian couples. Approximately, 20% of infertile couples are diagnosed with unexplained infertility and left without an explanation for their inability to have a baby. Pathological uterine receptivity and embryo implantation are hypothesized mechanisms underlying sub-fertility in these couples. Embryo implantation requires a complicated sequence of events involving the differentiation of endometrial cells to attain uterine receptivity and the synchronized interaction between maternal and embryonic tissues. Vitamin D has been hypothesized to play a role in this poorly understood process. Vitamin D is a known regulator of signal transduction pathways involved in embryo implantation and its receptors are involved in calcium-regulation in various reproductive tissues including, the ovary, uterus, and placenta. In Canada, the prevalence of Vitamin D insufficiency is approximately 34-50%. The goal of the proposed study is to determine the prevalence of vitamin D insufficiency in an infertile population and whether this prevalence is higher than in average Canadian reproductive age women. More importantly, we will investigate whether vitamin D insufficiency in our infertile population translates to impaired implantation and reduced clinical pregnancy rates. Insight into vitamin D's role in reproduction is essential not only to provide scientific understanding of the mechanism underlying embryo implantation, but also because vitamin D supplementation could provide an easy and safe means of treating infertility.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, < 40
* Day 3 FSH < 10
* Capable of providing informed consent

Exclusion Criteria:

* BMI > 35
* Untreated uterine pathology ie. fibroids, septum, polyps
* Unable to provide informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing IVF at Mount Sinai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
implantation rates following IVF | 3 weeks

SECONDARY OUTCOMES:
clinical pregnancy rates following IVF | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Liu, MD FRCSC, Principal Investigator — Mount Sinai Hospital, University of Toronto
Locations (1):
- Centre for Fertility and Reproductive Health, Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Garbedian K, Boggild M, Moody J, Liu KE. Effect of vitamin D status on clinical pregnancy rates following in vitro fertilization. CMAJ Open. 2013 Jun 28;1(2):E77-82. doi: 10.9778/cmajo.20120032. eCollection 2013 May. PMID 25077107